CLINICAL TRIAL: NCT00182429
Title: Prospective, Randomized Study of Oral Metronidazole vs. Oral Metronidazole and Rifampin for Treatment of Clostridium Difficile-associated Diarrhea (CDAD)
Brief Title: Efficacy of Metronidazole Versus Metronidazole and Rifampin in CDAD Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2261; Grant Number R03-39 (PSI)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Clostridium Enterocolitis; Antibiotic-Associated Diarrhea; Pseudomembranous Colitis; Pseudomembranous Enterocolitis; Pseudomembranous Enteritis
Keywords: Antibiotic associated diarrhea; C. difficile; Metronidazole; Rifampin
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — Metronidazole; Rifampin

INTERVENTIONS:
Drug: Metronidazole and Rifampin

SUMMARY:
What is the difference between the use of one drug (Oral Metronidazole) versus the use of this same drug combined with another drug (Rifampin) in treatment of bacteria and infection-associated diarrhea in patients? This infection is an important cause of morbidity and mortality in both the community and hospitals, and the leading cause of hospital and chronic facility-acquired diarrhea. Research is important for the treatment of this infection. Patient care with use of two medication treatment regimens will be studied.

DETAILED DESCRIPTION:
Clostridium difficile infection contributes to both community and hospital acquired morbidity and mortality. Metronidazole alone is usually considered the drug of choice, however, frequent relapses occur at a rate of 10-40%. The purpose of this study is to address the use of a combined drug regimen treatment (Metronidazole and Rifampin) for the treatment of CDAD. These drugs used together have been successful. Objectives are to determine the time (days) to resolution of symptoms in each treatment arm; to measure clinical relapse rates; and to assess adverse reactions related to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients + outpatients diagnosed with CDAD based on SHEA definition [Laboratory confirmation for presence of C.difficile toxin using enzyme immunoassay and no other etiology for diarrhea + Presence of 1 or more of the following: diarrhea (6 watery stool over 36 hours or 3 unformed stools in 24 hours for at least 2days), pseudomembranes at endoscopy].

Exclusion Criteria:

* Age < 14 yr
* Known hypersensitivity to metronidazole, rifampin
* Receiving medication(s) with potential significant drug interaction with rifampin
* Active liver disease as indicated by ALT > 200 U/L
* Adynamic ileus
* Toxic megacolon
* Pregnancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2004-02; Primary Completion 2005-04-30 (Actual); Study Completion 2005-12-31 (Actual)

PRIMARY OUTCOMES:
Resolution of symptoms in each treatment arm (in days) up to 40 days (measured using daily stool and symptom diary).

SECONDARY OUTCOMES:
Clinical relapse rate in each group (time to relapse in days) up to 40 days after initial diagnosis (measured by repeating C. difficile toxin assay and analyzing daily stool and symptom diary).
Adverse reactions related to treatment within 40 days (measured using daily symptom diary and interviewing patient).
Occurrance of metronidazole resistance in the organism (C. difficile) in relapse cases.

CONTACTS AND LOCATIONS:
Overall Officials: Christine H Lee, MD, Study Director — McMaster University
Locations (4):
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Henderson General Hospital, Hamilton, Ontario

REFERENCES:
- [Background] Buggy BP, Fekety R, Silva J Jr. Therapy of relapsing Clostridium difficile-associated diarrhea and colitis with the combination of vancomycin and rifampin. J Clin Gastroenterol. 1987 Apr;9(2):155-9. doi: 10.1097/00004836-198704000-00009. PMID 3571889
- [Background] Wenisch C, Parschalk B, Hasenhundl M, Hirschl AM, Graninger W. Comparison of vancomycin, teicoplanin, metronidazole, and fusidic acid for the treatment of Clostridium difficile-associated diarrhea. Clin Infect Dis. 1996 May;22(5):813-8. doi: 10.1093/clinids/22.5.813. PMID 8722937
- [Background] Young GP, Ward PB, Bayley N, Gordon D, Higgins G, Trapani JA, McDonald MI, Labrooy J, Hecker R. Antibiotic-associated colitis due to Clostridium difficile: double-blind comparison of vancomycin with bacitracin. Gastroenterology. 1985 Nov;89(5):1038-45. doi: 10.1016/0016-5085(85)90206-9. PMID 4043661
- [Background] Olson MM, Shanholtzer CJ, Lee JT Jr, Gerding DN. Ten years of prospective Clostridium difficile-associated disease surveillance and treatment at the Minneapolis VA Medical Center, 1982-1991. Infect Control Hosp Epidemiol. 1994 Jun;15(6):371-81. doi: 10.1086/646934. PMID 7632199
- [Background] Dudley MN, McLaughlin JC, Carrington G, Frick J, Nightingale CH, Quintiliani R. Oral bacitracin vs vancomycin therapy for Clostridium difficile-induced diarrhea. A randomized double-blind trial. Arch Intern Med. 1986 Jun;146(6):1101-4. PMID 3521518
- [Background] Teasley DG, Gerding DN, Olson MM, Peterson LR, Gebhard RL, Schwartz MJ, Lee JT Jr. Prospective randomised trial of metronidazole versus vancomycin for Clostridium-difficile-associated diarrhoea and colitis. Lancet. 1983 Nov 5;2(8358):1043-6. doi: 10.1016/s0140-6736(83)91036-x. PMID 6138597
- [Background] Barbut F, Decre D, Burghoffer B, Lesage D, Delisle F, Lalande V, Delmee M, Avesani V, Sano N, Coudert C, Petit JC. Antimicrobial susceptibilities and serogroups of clinical strains of Clostridium difficile isolated in France in 1991 and 1997. Antimicrob Agents Chemother. 1999 Nov;43(11):2607-11. doi: 10.1128/AAC.43.11.2607. PMID 10543736
- [Background] de Lalla F, Nicolin R, Rinaldi E, Scarpellini P, Rigoli R, Manfrin V, Tramarin A. Prospective study of oral teicoplanin versus oral vancomycin for therapy of pseudomembranous colitis and Clostridium difficile-associated diarrhea. Antimicrob Agents Chemother. 1992 Oct;36(10):2192-6. doi: 10.1128/AAC.36.10.2192. PMID 1444298